CLINICAL TRIAL: NCT07150429
Title: EVALUATION OF THE EFFECTIVENESS OF POSITIVE AND NEGATIVE VISUAL MATERIALS USED AS MOTIVATIONAL TOOLS IN ORAL HYGIENE EDUCATION ON CHILDREN'S ORAL HYGIENE PERFORMANCE
Brief Title: Impact of Visual Stimuli on Pediatric Oral Hygiene Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Merve CANDAN, Associate Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ESOGU-PEDO-05.06.2024/36
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dental Plaque; Halitosis; Oral Hygiene Education Methods
Keywords: dental plaque; halitosis; oral hygiene education; behavioral motivation
MeSH Terms: conditions — Dental Plaque; Halitosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verbal-active education supported by positive visual aids (Experimental)
  Interventions: Other: Verbal-Active Oral Hygiene Education with Positive Visual Aids
- Verbal-active education supported by negative visual aids (Experimental)
  Interventions: Other: Verbal-Active Oral Hygiene Education with Negative Visual Aids
- Verbal-active education only (control group) (Experimental)
  Interventions: Other: Verbal-Active Oral Hygiene Education (Control Group)

INTERVENTIONS:
Other: Verbal-Active Oral Hygiene Education with Negative Visual Aids — Verbal-Active Oral Hygiene Education with Visual Aid Variations
  Arms: Verbal-active education supported by negative visual aids
Other: Verbal-Active Oral Hygiene Education (Control Group) — Control group
  Arms: Verbal-active education only (control group)
Other: Verbal-Active Oral Hygiene Education with Positive Visual Aids — Verbal-Active Oral Hygiene Education with Visual Aid Variations
  Arms: Verbal-active education supported by positive visual aids

SUMMARY:
In the present study, children aged 7 to 14 will receive verbal and active (hands-on) oral hygiene education. The education will be delivered in three different formats:

Education supported with positive visual aids (images of healthy teeth),

Education supported with negative visual aids (images of decayed or unhealthy teeth),

Verbal and active education only (control group).

These visual aids are intended to demonstrate the potential positive and negative outcomes of tooth brushing behavior.

The aim of the study is to evaluate the effect of these different visual motivational tools approaches on children's oral hygiene performance.

To achieve this, the children's dental plaque levels and halitosis scores will be measured before the education, one week after, and one month after. These procedures are quick, painless, and non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* (1) children who had not previously received oral hygiene education, (2) children with carious lesions scored no higher than 4 on the ICDAS scale, and (3) systemically healthy children between the ages of 7 and 14. The study population consisted of male children, as well as female children who had not yet reached menarche.

Exclusion Criteria:

* (1) Children who declined to participate in the study, (2) girls who had reached menarche, (3)children with systemic disorders, and (4) children with presenting with intraoral conditions such as defective restorations that could facilitate plaque retention.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Dental plaque score | From baseline to 1st week and 1st month after the treatment
  Dental plaque score measured by Silness-Löe Index
Halitosis score | From baseline to 1st week and 1st month after the treatment
  Halitosis score assessment using the Rosenberg Organoleptic Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University Faculty of Dentistry Department of Pedodontics, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No